CLINICAL TRIAL: NCT00741650
Title: Ibedrift- Health Related Coping. A Randomized Controlled Trial Comparing a Worksite Educational Intervention With or Without Referral to Treatment as Usual.
Brief Title: Ibedrift- A Trial Comparing a New Approach to Musculoskeletal Pain Consisting of Education and Peer Involvement to Treatment as Usual
Acronym: Ibedrift
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: NORCE Norwegian Research Centre AS (Other)
Collaborators: Sykehuset i Vestfold HF (Other); Helse Sor-Ost (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 801622-611704; 18997 (Other: NSD); S-08054b (Other: REK)
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Neck Pain Musculoskeletal; Back Pain Lower Back
Keywords: Musculoskeletal pain; Brief cognitive intervention; Cognitive behavior therapy; Intervention Study; Health prevention; workplace intervention
MeSH Terms: conditions — Low Back Pain; Musculoskeletal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Information and peer advisor
  Interventions: Behavioral: Information and Peer advisor
- 2 (Experimental): Information, peer advisor and referral to further treatment
  Interventions: Behavioral: Information, peer advisor and fast referral
- 3 (No Intervention): Treatment as usual

INTERVENTIONS:
Behavioral: Information and Peer advisor — Information at work place and recruitment and training of one employee as a peer advisor who help colleagues who experience musculoskeletal pain with reasons to stay active, help with adjustment in the work situation to allow individuals to stay at work.
  Arms: 1
Behavioral: Information, peer advisor and fast referral — Information at work place and recruitment and training of one employee as a peer advisor who help colleagues who experience musculoskeletal pain with reasons to stay active, help with adjustment in the work situation to allow individuals to stay at work.
  In addition, the peer advisor can refer employees who do not improve to a two day educational program that also includes a medical exam and individual counselling.
  In addition,
  Arms: 2

SUMMARY:
A randomized controlled trial comparing a new approach to musculoskeletal pain consisting of education and peer involvement to treatment as usual. All local government employees in 1-3 Norwegian municipalities will be invited to participate.

DETAILED DESCRIPTION:
The purpose of the study is to systematically test a new treatment method for musculoskeletal pain in Norway. The intervention focuses on attempting to treat musculoskeletal pain outside the traditional medical system as much as possible, to avoid the establishment of a patient identity and passive patient behavior. In addition, participants are given reasons to stay active, and not advice to stay active.

Ibedrift is a randomized controlled trial with the aim of studying the effect of a new treatment regime for musculoskeletal pain, focusing on didactic information about low back pain with peer support. Those participants not in the control group will have the option of contacting a peer advisor, a non health professional trained by the iBedrift crew to give information about back pain and reasons to stay active. For those who have not recovered within a short period of time, and who are randomized to full treatment, the peer advisor can send them directly to health personnel for a brief intervention consisting of a medical examination with screening for conditions that need treatment, counseling and education.

The intervention was done in 2 Norwegian municipalities for all local government employees. Randomization was done at the level of working units (schools, offices etc) which allows for more message containment.

ELIGIBILITY:
Inclusion Criteria:

* All employees above 18 years

Exclusion Criteria:

* Cancer
* Known congenital musculoskeletal disease
* Cauda equina syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2097 (Actual)
Dates: Start 2008-09; Primary Completion 2011-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Sick Leave | 1 year and 2 year after start of intervention

SECONDARY OUTCOMES:
Low Back pain | 1 year and 2 years after intervention
Subjective Health complaints | 1 year and 2 years after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Aage Indahl, Ph.d, Principal Investigator — The Hospital of Vestfold
Locations (1):
- Spesialsykehuset for Rehabilitering, Stavern, Norway

REFERENCES:
- [Background] Odeen M, Ihlebaek C, Indahl A, Wormgoor ME, Lie SA, Eriksen HR. Effect of peer-based low back pain information and reassurance at the workplace on sick leave: a cluster randomized trial. J Occup Rehabil. 2013 Jun;23(2):209-19. doi: 10.1007/s10926-013-9451-z. PMID 23657490
- [Background] Ree E, Odeen M, Eriksen HR, Indahl A, Ihlebaek C, Hetland J, Harris A. Subjective health complaints and self-rated health: are expectancies more important than socioeconomic status and workload? Int J Behav Med. 2014 Jun;21(3):411-20. doi: 10.1007/s12529-013-9329-7. PMID 23868103